CLINICAL TRIAL: NCT03727087
Title: Blood Sample Collection to Evaluate Biomarkers in Subjects With Untreated Melanoma
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-03
Record Dates: First submitted 2018-10-23; First posted 2018-11-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Melanoma: Subjects with clinically confirmed melanoma or high suspicion of a primary malignancy of melanoma based on skin exam or imaging and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment.

SUMMARY:
The primary objective of this study is to obtain de-identified, clinically characterized, whole blood specimens to evaluate biomarkers associated with cancer for diagnostic assay development.

DETAILED DESCRIPTION:
Subjects will have been recently diagnosed with untreated melanoma. Subjects will have a blood sample collected at enrollment and provide medical history prior to initiation of treatment. There will be no further follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female > 18 years of age.
2. Subject has an untreated primary melanoma.

   OR

   Subject has high suspicion of primary malignancy of melanoma based on skin exam or imaging.
3. Subject understands the study procedures and is able to provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Any previous cancer diagnosis within the past 5 years (with the exceptions of basal cell or squamous cell skin cancers).
2. Chemotherapy and/or radiation therapy within 5 years prior to enrollment/sample collection.
3. Any treatment for the primary malignancy or sites of metastases. Subject may not have started neo-adjuvant chemotherapy, neo-adjuvant radiation therapy, immunotherapy or other treatment and/or surgery prior to blood sample collection.
4. Less than 3 days between fine needle aspiration (FNA) of target pathology and blood collection.
5. Less than 5 days between biopsy (other than FNA) of target pathology and blood collection.
6. IV contrast (e.g. CT and MRI) within 1 day [or 24 hours] of blood collection.
7. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 350 subjects will be enrolled. Subjects will be men and women, 18 years of age and older, who have an untreated melanoma or a high suspicion of primary malignancy of melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Blood-based biomarkers associated with genetic and epigenetic alterations. | Point in time blood collection (1 day) at enrollment
  Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in blood from subjects with melanoma at the pre-intervention stage.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - CARTI Cancer Center, Little Rock, Arkansas
  - Alliance Research Centers, Laguna Hills, California
  - Palmtree Clinical Research, Inc, Palm Springs, California
  - San Fernando Valley Health Institute, Van Nuys, California
  - Middlesex Hospital, Middletown, Connecticut
  - The Stamford Hospital, Stamford, Connecticut
  - Direct Helpers Research Center, Hialeah, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Mid-Florida Hematology and Oncology Center, Orange City, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Balanced Life Health Care Solutions, LLC, Buford, Georgia
  - IACT Health (DBA John B. Amos Cancer Center), Columbus, Georgia
  - PMG Research, INC, Downers Grove, Illinois
  - Carle Cancer Center NCI, Urbana, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - DermAssociates, PC, Rockville, Maryland
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - HealthPartner Institute, Bloomington, Minnesota
  - MediSync Clinical Research, Petal, Mississippi
  - Somnos Laboratories, Inc., Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - East Carolina University Brody School of Medicine, Greenville, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - MediSync Clinical Research, Dayton, Ohio
  - Spartanburg Regional Healthcare District, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - The Jackson Clinic Professional Association, Jackson, Tennessee
  - MediSync Clinical Research, Austin, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - MediSync Clinical Research, Pflugerville, Texas
  - Aim Trials, LLC, Plano, Texas
  - Wenatchee Valley Hospital, Wenatchee, Washington
  - Dean Clinic - Fort Atkinson Specialty Services, Fort Atkinson, Wisconsin
  - HSHS St Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - ProHealth Care, Oconomowoc, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol and informed consent form (when applicable) will also be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.